CLINICAL TRIAL: NCT00764270
Title: The Role of R-alpha Lipoic Acid in the Treatment of Atherosclerotic Vascular Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Oregon Health and Science University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gerd Bobe, Principal Investigator, Linus Pauling Institute Associate Professor, Department of Animal and Rangeland Sciences, Oregon State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT002034-2 (7187); 5P01AT002034 (NIH)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; lipoic acid; thioctic acid; triglycerides; overweight; obesity; oxidative stress; inflammation
MeSH Terms: conditions — Atherosclerosis; Overweight; Obesity; Inflammation | interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: Crossover study in which participants are randomly assigned to the sequence of receiving R-Alpha Lipoic Acid and Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipoic acid treatment (Active Comparator): Participants take lipoic acid with a washout period before or after placebo.
  Interventions: Dietary Supplement: R-alpha lipoic acid
- Placebo treatment (Placebo Comparator): Participants take placebo with a washout period before or after lipoic acid treatment
  Interventions: Dietary Supplement: R-alpha lipoic acid

INTERVENTIONS:
Dietary Supplement: R-alpha lipoic acid — 300 mg R-alpha lipoic acid or placebo twice daily for 12 weeks, followed by a washout period of 12 weeks, followed by another treatment phase of the other treatment placebo or 300 mg R-alpha-lipoic acid for 12 weeks

SUMMARY:
The purpose of this study is to see if a dietary supplement, R-alpha lipoic acid, is able to reduce risk factors in people with documented heart disease and increased levels of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Documented congestive heart disease (CHD)(defined as at least one significant coronary stenosis > 50% on angiography, or history of documented myocardial infarction)
* Not diagnosed with unstable angina, uncontrolled hypertension, heart failure, recent myocardial infarction (within last six months)
* Not taking insulin or oral hypoglycemic agents, anti-inflammatory drugs other than aspirin, or hormone replacement therapy
* On stable doses for four weeks prior to entry of lipid-lowering therapy (statins), aspirin, and angiotensin-converting enzyme inhibitors or other blood pressure medications. P
* No tobacco use within 3 months of the study
* No laboratory evidence of renal, hepatic, or hematological abnormalities
* Not currently taking vitamin or antioxidant supplements, including R-alpha lipoic acid, except standard multivitamin/mineral supplements containing not more than the Daily Value (DV) of the vitamins and minerals;
* Elevated levels of urinary and plasma F2-isoprostanes
* Elevated plasma levels of hs-CRP

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
hs-CRP | 12,20 & 32 weeks
  High sensitive C-reactive protein

SECONDARY OUTCOMES:
8-lso-PGF2a | 12, 20 & 32 weeks
  8-iso-prostaglandin F2alpha

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Bobe, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States